CLINICAL TRIAL: NCT01689766
Title: A Screening Study Using FolateScan to Identify Subjects With Folate Receptor-Positive Metastatic Renal Cell Carcinoma
Brief Title: Study Using FolateScan to Identify Subjects With Folate Receptor-Positive Metastatic Renal Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Endocyte (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: EC20.9
Record Dates: First submitted 2012-09-09; First posted 2012-09-21 (Estimated); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Metastatic Renal Cell Carcinoma
Keywords: Renal Cell
MeSH Terms: conditions — Carcinoma, Renal Cell

ARMS (1):
- Technetium Tc 99m EC20 (Other)
  Interventions: Drug: Technetium Tc 99m EC20

INTERVENTIONS:
Drug: Technetium Tc 99m EC20

SUMMARY:
Phase 2, multi-center, open-label, single-treatment group, baseline-controlled study to identify subjects with Folate Receptor-Positive Metastatic Renal Cell Carcinoma

DETAILED DESCRIPTION:
The investigational new drug (FolateScan or Technetium Tc 99m EC20) is a folate-targeted diagnostic radiopharmaceutical agent designed to bind to the folate receptor. The folate receptor is a glycoprotein that is over-expressed in many types of cancer cells but it is only minimally distributed in normal tissues . Folate conjugates bind to the folate receptor with high affinity and are brought into the cell via endocytosis. In contrast, folic acid itself enters most normal cells via the reduced folate carrier, a pathway entirely inaccessible to folate conjugates. Therefore, these folate conjugates are specific to cancer cells.

This is a phase 2, multi-center, open-label, single-treatment group, baseline-controlled study designed to verify product safety, gather data on the percentage of metastatic renal cell carcinoma patients with increased uptake of FolateScan in tumors, and to calculate sensitivity, specificity, accuracy, positive predictive value, and negative predictive value of FolateScan compared to immunohistochemical staining (IHC).

ELIGIBILITY:
Inclusion Criteria:

* To be eligible for the study, patients must fulfill all of the following criteria:

  1. Patient must be 18 years of age or older.
  2. Patient must have suspected metastatic renal cell carcinoma with at least one identifiable lesion >2.0 cm as diagnosed by CT, MRI, or ultrasonography within 60 days prior to enrollment.
  3. Patient must have good kidney function defined as a serum creatinine ≤1.5 X ULN.
  4. Patient must provide written informed consent prior to enrollment.
  5. Patients must provide a formalin-fixed, paraffin-embedded tissue sample of either the primary or metastatic or recurrent site(s) for IHC staining for the presence of folate receptors from either a previous surgical/biopsy procedure or from a surgery/biopsy scheduled within 30 days of FolateScan. A fine needle aspirate is not acceptable.

Exclusion Criteria:

* Any of the following criteria will make the patient ineligible to participate in this study:

  1. Patient is pregnant or breastfeeding.
  2. Patient is simultaneously participating in another investigational drug study, excluding the follow-up phase.
  3. Patient has received an investigational agent or therapeutic chemotherapy within 7 days prior to enrollment.
  4. Patient is unable to tolerate conditions for radionuclide imaging.
  5. Patient has been administered another radiopharmaceutical that would interfere with the assessment of Technetium Tc 99m EC20.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2003-11; Primary Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Mayo Clinic, Rochester, Minnesota
  - Baylor College of Medicine, Houston, Texas